CLINICAL TRIAL: NCT03021733
Title: A Pilot Cohort Study of Surgical and Non-surgical Management of Rotator Cuff Tears
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Joel Gagnier, Assistant Professor, University of Michigan
Other Study IDs: HUM00056320
Record Dates: First submitted 2017-01-12; First posted 2017-01-16 (Estimated); Last update posted 2017-09-18 (Actual); Status verified 2017-09

CONDITIONS: Full Thickness Rotator Cuff Tear

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Non-operative: Patients whom elected non-operative treatment
- Operative: Patients whom elected operative treatment
  Interventions: Procedure: Operative management

INTERVENTIONS:
Procedure: Operative management — Rotator cuff surgery
  Groups: Operative

SUMMARY:
This project will involve planning and implementing a two-arm prospective pragmatic cohort clinical trial in patients with known rotator cuff tears.

DETAILED DESCRIPTION:
This project will involve planning and implementing a two-arm prospective pragmatic cohort clinical trial in patients with known rotator cuff tears. Pragmatic or effectiveness clinical trials reflect real world settings and thus have greater external generalizability than efficacy trials. The evaluation component in this trial will be three-fold: first, the study team will compare the success of patients undergoing operative versus non-operative management and identify which variables predict success in each group; second, investigators will attempt to predict which patients end up choosing, along with their care giver(s), operative versus non-operative management by examining the predictive capability of a selection of variables; third, investigators will evaluate the clinical research site(s), personnel, and implementation processes for their capability to implement clinical trials with the intent of planning for a future large multi-site clinical trial building on the results of the present study.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age with full-thickness rotator cuff tears eligible for operative repair

Exclusion Criteria:

* less than 18 years old,
* non-operative rotator cuff tears,
* calcific tendonitis, fracture, adhesive capsulitis,
* severe osteoarthritis of the shoulder,
* no prior shoulder surgery

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients presenting to an orthopaedic clinic with full-thickness rotator cuff tears as determined by surgeon opinion and imaging
Sampling Method: Non-Probability Sample
Enrollment: 222 (Actual)
Dates: Start 2012-02; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Veterans Rand VR-12 Quality of Life Score | baseline
Veterans Rand VR-12 Quality of Life Score | 4 weeks
Veterans Rand VR-12 Quality of Life Score | 8 weeks
Veterans Rand VR-12 Quality of Life Score | 16 weeks
Veterans Rand VR-12 Quality of Life Score | 32 weeks
Veterans Rand VR-12 Quality of Life Score | 48 weeks
Veterans Rand VR-12 Quality of Life Score | 64 weeks

IPD SHARING:
Plan to Share IPD: No
No individual patient data will be shared